CLINICAL TRIAL: NCT02448290
Title: Phase II, Single-arm Study of Selumetinib in Combination With Docetaxel, in Advanced Gastric Adenocarcinoma Patients With Low/High MEK Signature, RAS Mutation or RAS Amplification as a Second-line Chemotherapy
Brief Title: Single-arm Study of Selumetinib in Combination With Docetaxel, in Advanced Gastric Adenocarcinoma Patients With Low/High MEK Signature, RAS Mutation or RAS Amplification as a Second-line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Division of Hematology-Oncology, Department of Medicine, Samsung Medical Center,, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-04-126
Record Dates: First submitted 2015-01-15; First posted 2015-05-19 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Gastric Adenocarcinoma
Keywords: gastric adenocarcinoma patients with low/high MEK signature,
MeSH Terms: interventions — Docetaxel; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel+selumetinib (Experimental): Selumetinib 75 mg will be administered orally twice a day with continuous dosing schedule Docetaxel 60 mg/m2 will be administered via intravenous access every 3 weeks.
  Interventions: Drug: docetaxel plus selumetinib

INTERVENTIONS:
Drug: docetaxel plus selumetinib — Selumetinib will be administered orally 75mg twice a day continuously. Docetaxel will be administered as an IV infusion over 1 hour at 60 mg/m2 every 3 week of a 21 days schedule.

SUMMARY:
This study is a single-arm, phase II study of selumetinib in combination with docetaxel in patients with advanced gastric adenocarcinoma harboring MEK signature, RAS mutation or amplification as a second line chemotherapy.

Selumetinib will be administered orally 75mg twice a day continuously. Docetaxel will be administered as an IV infusion over 1 hour at 60 mg/m2 every 3 week of a 21 days schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after firstline therapy.

   * The 1st line regimen must have contained doublet 5-fluoropyrimidine and platinum based regimen.
   * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doublet 5-fluoropyrimidine and platinum-based regimen could be considered as 1st line therapy.
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the 1st line therapy.
5. Provision of tumor sample (from either a resection or biopsy)
6. Patients with MEK signature, RAS mutation or amplification through the VIKTORY trial.

   (The VIKTORY trial uses Ion Torrent PGM to screen for a panel of cancer mutations and nanostring, copy number variation panel (see addendum for the VIKTORY trial)
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
8. ECOG performance status 0-1.
9. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
10. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥9.0 g/L (transfusion allowed)
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * White blood cells (WBC) > 3 x 109/L
    * Platelet count ≥100 x 109/L (transfusion allowed)
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (does not include patients with Glibert's disease)
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
    * Serum creatinine ≤1.5 x institutional ULN
11. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
12. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. for women of childbearing potential.
13. Provision of consent for mandatory biopsy at progression

Exclusion Criteria:

1. More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.
2. Any previous treatment with MEK, RAS or RAF inhibitors
3. Any previous treatment with docetaxel.
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
5. HER2 positive patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)
6. Patients unable to swallow orally administered medication.
7. Treatment with any investigational product during the last 14 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
8. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denusomab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
9. Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.
10. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
11. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
12. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
13. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Baseline Left ventricular ejection fraction below the LLN of <55% measured by echocardiography or institution's LLN for MUGA, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
14. Ophthalmological conditions as follows:Intra-ocular pressure >21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure), Current or past history of retinal pigment epithelial detachment/central serous retinopathy or or current or past history retinal vein occlusion
15. Female patients who are breast-feeding or child-bearing and Male or female patients of reproductive potential who are not employing an effective method of contraception
16. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
response rate | 24 weeks

SECONDARY OUTCOMES:
duration of response | 24 weeks
disease control rate | 8weeks
overall survival | up to 100weeks
progression-free survival | up to 100weeks
safety assessed by safety( AEs/SAEs) | up to 100weeks
  The following parameters will be recorded for each ECG: date and time of ECG, heart rate (beats/min), QT (ms), QTcB (ms), sinus rhythm (yes/no), and overall evaluation (normal/abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, MD, PhD, Principal Investigator — Division of Hematology-Oncology, Department of Medicine, Samsung Medical Center,
Locations (1):
- Samsung Medical center, Seoul, South Korea